CLINICAL TRIAL: NCT00947336
Title: Evaluation of Safety and Efficacy of Synbiotic on the Incidence and Recurrence of Spontaneous Bacterial Peritonitis in Cirrhotics: A Randomized, Double Blind Placebo Controlled Trial
Brief Title: Evaluation of Safety & Efficacy of Synbiotic on the Incidence and Recurrence of Spontaneous Bacterial Peritonitis (SBP) in Cirrhotics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Collaborators: Jhaver Research Foundation Limited (Unknown)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 2009-PHT-01
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2009-07

CONDITIONS: Cirrhosis With Ascites
MeSH Terms: interventions — Norfloxacin; Synbiotics

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Norfloxacin + Synbiotic (Active Comparator)
  Interventions: Drug: Norfloxacin + Synbiotic
- Norfloxacin + Placebo (Placebo Comparator)
  Interventions: Drug: Norfloxacin + Placebo

INTERVENTIONS:
Drug: Norfloxacin + Synbiotic — Norfloxacin 400 mg once daily with synbiotic capsules (Streptococcus faecalis JPC 30 million, Clostridium butyricum 2 million, Bacillus mesentericus JPC 1 million, Lactobacillus sporogenes 50 million spores) 2 t.i.d.
  Arms: Norfloxacin + Synbiotic
Drug: Norfloxacin + Placebo — Norfloxacin 400 mg once daily with placebo
  Arms: Norfloxacin + Placebo

SUMMARY:
Background: Spontaneous bacterial peritonitis (SBP) is a serious complication in patients of cirrhosis with ascites and may occur despite antibiotic prophylaxis. Small bowel dysmotility and bacterial overgrowth have been documented to be related to SBP. Aims: To investigate whether addition of prebiotic plus probiotics (synbiotics) to norfloxacin enhances the efficacy of norfloxacin in prevention of SBP in high risk patients with ascites.

Methods: A prospective, double blind, randomized controlled trial was conducted in consecutive high-risk cirrhotic patients with ascites who had either recovered from an episode of SBP (secondary prophylaxis) or who never had SBP but were at high risk for development of SBP (low ascitic fluid protein or serum bilirubin ≥2.5 mg/dL; primary prophylaxis). Norfloxacin 400 mg once daily with synbiotic capsules (Streptococcus faecalis JPC 30 million, Clostridium butyricum 2 million, Bacillus mesentericus JPC 1 million, Lactobacillus sporogenes 50 million spores) 2 t.i.d. (group I) or norfloxacin 400 mg once daily with placebo (group II) was given and occurrence of SBP within a period of 6 months (primary endpoint) or side-effects of therapy and mortality (secondary endpoints) were recorded. Every patient received IV albumin to maintain a serum albumin level of >3.2 g/dl. SBP was treated with intravenous antibiotics with albumin.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis with ascites with any one of following:

  * History of at least one episode of SBP, or
  * Ascitic fluid protein less than or equal to 1g/dL, or
  * Serum bilirubin more than or equal to 2.5 mg/dL

Exclusion Criteria:

* Renal failure
* HCC
* Hepatic encephalopathy
* No consent

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2005-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Development of SBP | 6 months

SECONDARY OUTCOMES:
Mortality | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, G B Pant Hospital, New Delhi, National Capital Territory of Delhi, India